CLINICAL TRIAL: NCT03640299
Title: Shanghai First Maternity and Infant Hospital
Brief Title: The Safety and Efficacy of Enhanced Recovery After Surgery on Clinical and Immune Outcomes for Gynecological Oncology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERAS GYNMT LSC
Record Dates: First submitted 2018-07-08; First posted 2018-08-21 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Gynecologic Cancer
Keywords: Gynecologic Cancer; Enhanced Recovery After Surgery; Laparoscopic surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS procedure (Experimental): In this arm, ERAS perioperative cares patients planned to undergoing laparoscopic surgery, following the ERAS protocols.
  Extensive preoperative counselling and education by surgeon and anesthetists.
  No Bowel preparation.
  6 h fast for solid food and carbohydrate loading with clear fuilds 2h before surgery.
  Oral nonselective NSAIDs premedication.
  Total Intravenous Anesthesia via TCI, wound infiltration and the transversus abdominis plane (TAP).
  Minimally invasive surgery.
  Maintenance of normothermia.
  Avoidance of surgical drains and nasogastric tubes.
  Nonselective NSAIDs postoperative medication.
  Postoperative nausea and vomiting active control.
  Early oral feeding and ambulation.
  VTE prophylaxis postoperative.
  Interventions: Procedure: ERAS procedure
- Traditional treatment procedure (No Intervention): In this arm, control patients planned to undergoing laparoscopic surgery, following the traditional treatment protocols.
  Conventional preoperative visits and education.
  Mechanical bowel preparation.
  Fasting overnight, and no fluids before surgery.
  No oral nonselective NSAIDs premedication.
  Continuous epidural anesthesia is administered before surgery. Sevoflurane and sufentanil maintain the depth of anesthesia.
  Minimally invasive surgery.
  No maintenance of normothermia.
  Drainage tube insertion if needed.
  Postoperative patient-controlled intravenous analgesia.
  Postoperative Nausea Control if needed.
  Conventional oral feeding and mobilization.
  No bowel routine.
  VTE prophylaxis postoperative.

INTERVENTIONS:
Procedure: ERAS procedure — Optimized preoperative, intraoperative and postoperative procedures.
  Arms: ERAS procedure

SUMMARY:
The aim of this study is to compare outcomes of enhanced recovery after surgery (ERAS) procedure, involving preoperative, intraoperative and postoperative optimization, with those of conventional treatment procedure in women undergoing laparoscopic surgery for gynecologic cancer or suspected gynecologic cancer. Investigators hypothesize that those patients randomized to the ERAS protocol will have better recovery status, shorter lengths of hospital stay, without increasing readmission rates and complications, compared with traditional treatment.

DETAILED DESCRIPTION:
Over the past two decades, enhanced recovery after surgery (ERAS) has been initiated and developed in colorectal surgery by Kehlet. Studies have demonstrated that ERAS program can reduce length of hospital stay, hospital cost, complications and morbidity and improve the quality of patient recovery in colorectal, urologic, thoracic, orthopedic, and vascular surgeries by randomized trials and meta-analyses. However, the data in gynecologic oncology underwent minimally invasive therapy is scarce. Therefore, the aim of this study is compare outcomes of ERAS procedure with conventional treatment procedure, to provide practical experience and guidance for the treatment of gynecologic cancer in the future.

The study is a single-center randomized control trial (RCT), and 80 cases of gynecological malignancy in Shanghai First Maternity and Infant Hospital from 2018 to 2021 will be enrolled in this research. All patients with a known or suspected gynecologic malignancy scheduled for laparoscopic surgery will be screened for study eligibility. Those eligible for the study will be approached for participation in the study and provided written informed consent. The randomization sequence of group allocation by means of computer-generated random numbers was generated by an independent statistician from Tongji University.

For ERAS group, patients would receive an optimized preoperative, intraoperative and postoperative care, including extensive preoperative counselling, no mechanical bowel preparation, nonselective NSAIDs premedication, no preoperative fasting but with preoperative carbohydrate loading, tailored anaesthesiology, non-opioid pain management, early removal of urinary catheter, early postoperative feeding and mobilization, and postoperative antiemetic and analgesia management. For control group, patients would receive standard conventional procedure. After meeting the discharge criteria, patients would discharge and additionally follow-up in gynecologic oncology clinic at 2 weeks and 6 weeks postoperatively.

Primary outcome measure of the study involves operation length(h), intraoperative blood loss(mL), intraoperative fluid transfusion units(mL), intraoperative urinary volume(mL), intraoperative blood transfusion(mL), postoperative vital signs, Visual Analog Score (VAS) scale, Post Operative Nausea And Vomiting (PONV) status, first exhaust defecation time, ambulation, length of stay, hospitalization expense, albumin and prealbumin, and postoperative complications. Apart from clinical outcomes, the immunological indicators will also be assessed, consist of WBC, neutrophil count (NEUT), C-Reactive Protein (CRP), CD3+ T cells, CD4+ T cells, CD8+ T cells, CD4+/CD8+ T cells preoperatively, and on post-operative day 1(POD1), POD3, POD5. In addition, the anxiety and sleep quality indicators were analyzed by questionnaire preoperatively and POD5.

For statistical analyses, categorical variables were described using counts and frequencies, and quantitative variables were described using mean, medians and ranges. Patients' characteristics and distribution were compared with MannWhitney U and χ2 tests. The level of statistical significance was set at P< 0.05. Statistical analyses were carried out with the SPSS 20.0.

ELIGIBILITY:
Inclusion Criteria:

Newly pathological diagnosed and suspected gynecologic tumors, including cervical cancer, ovarian cancer, endometrial cancer, fallopian tube cancer, uterine carcinosarcoma, and choriocarcinoma.

Ages range from 18 to 70.

body mass index of between 18 and 35.

American Society of Anesthesiologists (ASA) grading of I to III.

No history of abdominal surgery and severe organ dysfunction such as heart and lung.

Exclusion Criteria:

Unwillingness to participate.

Inability to give written informed consent.

Absolute contraindication for surgery.

History of other malignancies, radiotherapy and chemotherapy.

Uncontrollable Cardiovascular and cerebrovascular diseases, diabetes, and liver and kidney dysfunction.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-08-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Total length of hospital stay (days) | Up to 20 days
  Total length of hospital stay (days)

SECONDARY OUTCOMES:
Operation Time(h) | The day of surgery
  Operation Time(h)
Intraoperative blood loss(mL) | The day of surgery
  Blood loss during the operation
Intraoperative fluid transfusion units(mL) | The day of surgery
  Fluid transfusion units during the operation
Intraoperative urinary volume(mL) | The day of surgery
  Urinary volume during the operation
Intraoperative blood transfusion(mL) | The day of surgery
  Urinary volume during the operation
Visual Analog Score (VAS) for pain | Up to 5 days after surgery
  Visual Analog Score (VAS) for pain
Post Operative Nausea And Vomiting (PONV) status | Up to 5 days after surgery
  Post Operative Nausea And Vomiting (PONV) status
Time of off-bed activity per day | 1 week
  Postoperative activity
Distance of off-bed activity per day | 1 week
  Postoperative activity
First exhaust defecation time | Up to 3 days after surgery
  Bowel function recovery
Albumin | Before the operation, on Postoperative Day 1, Postoperative Day 3 and Postoperative Day 5
  Nutritional indicators
Prealbumin | Before the operation, on Postoperative Day 1, Postoperative Day 3 and Postoperative Day 5
  Nutritional indicators
WBC | Before the operation, on Postoperative Day 1, Postoperative Day 3 and Postoperative Day 5
  Immunological indicators
Neutrophil count (NEUT) | Before the operation, on Postoperative Day 1, Postoperative Day 3 and Postoperative Day 5
  Immunological indicators
C-Reactive Protein (CRP) | Before the operation, on Postoperative Day 1, Postoperative Day 3 and Postoperative Day 5
  Immunological indicators
CD4+ | Before the operation, on Postoperative Day 1, Postoperative Day 3 and Postoperative Day 5
  Immunological indicators
CD8+ | Before the operation, on Postoperative Day 1, Postoperative Day 3 and Postoperative Day 5
  Immunological indicators
CD4+ / CD8+ | Before the operation, on Postoperative Day 1, Postoperative Day 3 and Postoperative Day 5
  Immunological indicators
Hospitalization Expense | Up to 1 month after surgery
  Medical expense
Anxiety indicators | Before the operation and Postoperative Day 5
  Anxiety index were tested by questionnaire of self-rating anxiety scale(SAS) on preoperation and Postoperative Day 5
Sleep quality indicators | Before the operation and Postoperative Day 5
  Sleep quality index were tested by questionnaire of Pittsburgh sleep quality index(PSQI) on preoperation and Postoperative Day 5
Postoperative complications | Up to 1 month after surgery
  Postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqing Guo, Docter, Principal Investigator — Shanghai First Maternity and Infant Hospital
Locations (1):
- Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kehlet H. Multimodal approach to control postoperative pathophysiology and rehabilitation. Br J Anaesth. 1997 May;78(5):606-17. doi: 10.1093/bja/78.5.606. PMID 9175983
- [Background] Ni TG, Yang HT, Zhang H, Meng HP, Li B. Enhanced recovery after surgery programs in patients undergoing hepatectomy: A meta-analysis. World J Gastroenterol. 2015 Aug 14;21(30):9209-16. doi: 10.3748/wjg.v21.i30.9209. PMID 26290648
- [Background] Vlug MS, Wind J, Hollmann MW, Ubbink DT, Cense HA, Engel AF, Gerhards MF, van Wagensveld BA, van der Zaag ES, van Geloven AA, Sprangers MA, Cuesta MA, Bemelman WA; LAFA study group. Laparoscopy in combination with fast track multimodal management is the best perioperative strategy in patients undergoing colonic surgery: a randomized clinical trial (LAFA-study). Ann Surg. 2011 Dec;254(6):868-75. doi: 10.1097/SLA.0b013e31821fd1ce. PMID 21597360
- [Background] Wainwright TW, Immins T, Middleton RG. Enhanced recovery after surgery (ERAS) and its applicability for major spine surgery. Best Pract Res Clin Anaesthesiol. 2016 Mar;30(1):91-102. doi: 10.1016/j.bpa.2015.11.001. Epub 2015 Nov 23. PMID 27036606
- [Background] Nelson G, Altman AD, Nick A, Meyer LA, Ramirez PT, Achtari C, Antrobus J, Huang J, Scott M, Wijk L, Acheson N, Ljungqvist O, Dowdy SC. Guidelines for pre- and intra-operative care in gynecologic/oncology surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations--Part I. Gynecol Oncol. 2016 Feb;140(2):313-22. doi: 10.1016/j.ygyno.2015.11.015. Epub 2015 Nov 18. No abstract available. PMID 26603969
- [Background] Nelson G, Altman AD, Nick A, Meyer LA, Ramirez PT, Achtari C, Antrobus J, Huang J, Scott M, Wijk L, Acheson N, Ljungqvist O, Dowdy SC. Guidelines for postoperative care in gynecologic/oncology surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations--Part II. Gynecol Oncol. 2016 Feb;140(2):323-32. doi: 10.1016/j.ygyno.2015.12.019. Epub 2016 Jan 3. No abstract available. PMID 26757238
- [Background] Nelson G, Dowdy SC, Lasala J, Mena G, Bakkum-Gamez J, Meyer LA, Iniesta MD, Ramirez PT. Enhanced recovery after surgery (ERAS(R)) in gynecologic oncology - Practical considerations for program development. Gynecol Oncol. 2017 Dec;147(3):617-620. doi: 10.1016/j.ygyno.2017.09.023. Epub 2017 Sep 23. No abstract available. PMID 28947172
- [Derived] Chau JPC, Liu X, Lo SHS, Chien WT, Hui SK, Choi KC, Zhao J. Perioperative enhanced recovery programmes for women with gynaecological cancers. Cochrane Database Syst Rev. 2022 Mar 15;3(3):CD008239. doi: 10.1002/14651858.CD008239.pub5. PMID 35289396